CLINICAL TRIAL: NCT04469426
Title: Interactive Online Informational and Peer Support App for Patients with Low Anterior Resection Syndrome (LARS): a Multicenter Randomized Controlled Trial
Brief Title: Interactive Online Informational and Peer Support App for Patients with Low Anterior Resection Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Providence Healthcare (Other); Mount Sinai Hospital, Canada (Other); University Health Network, Toronto (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Assistant Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JGH-2020-2073
Record Dates: First submitted 2020-03-23; First posted 2020-07-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Patient Empowerment; Low Anterior Resection Syndrome; Colo-rectal Cancer; Peer Group; Patient Satisfaction; Health Attitude; Health Knowledge, Attitudes, Practice
Keywords: colorectal surgery; peer support
MeSH Terms: conditions — Patient Participation; Low Anterior Resection Syndrome; Colonic Neoplasms; Patient Satisfaction; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Informational online app group (Experimental): Participants will have access to an interactive online peer support app developed by the research team.
  Interventions: Other: Interactive online informational and peer support app
- Booklet only (No Intervention): Participants will only have access to the educational booklet on LARS developed by the colorectal research team.

INTERVENTIONS:
Other: Interactive online informational and peer support app — The app contains LARS information, bowel function diaries, and online platform with trained peer support mentor
  Arms: Informational online app group

SUMMARY:
After surgery for rectal cancer, many people undergo changes in bowel habits, which may include the need to empty their bowels more often, accidental leakage of stool or gas, the sudden urge to go to the bathroom, and more. The term "Low Anterior Resection Syndrome" or LARS is used to describe these symptoms. LARS has a negative impact on one's quality of life, and can lead to frustration, as there is no single intervention that has proven to be effective for LARS, and each patient has to undergo trial and error to find one's solution. As people struggle with LARS, they describe feeling hopeless and isolated. Peer support is a supportive relationship between individuals who share common experiences or face similar challenges. The goal of our study is to evaluate whether use of an online peer support application with trained mentors who themselves have lived or are living with LARS will empower patients to better manage their LARS symptoms and improve their quality of life.

DETAILED DESCRIPTION:
Restorative proctectomy is increasingly being performed for rectal cancer, allowing patients to avoid permanent colostomy. Low Anterior Resection Syndrome (LARS) refers to a constellation of bowel symptoms including frequency, urgency, incontinence, and clustering of bowel movements, that can affect up to 70 to 90% of patients following restorative proctectomy. Symptoms can last up to 15 years after resection. Currently, there is no standard treatment for LARS and management is symptom-based and reactive, rather than proactive. A recent focus group conducted at our institution among LARS patients and caregivers showed that people living with LARS experience anxiety and isolation due to their symptoms.

Peer support could be an important psychosocial intervention for people living with LARS, helping them normalize and validate their experience. Peer support refers to a supportive relationship between individuals who share common experiences or face similar challenges. This approach has been associated with positive physical and mental health outcomes for several patient populations. Our research group conducted a comprehensive review of online health information for patients with LARS, and demonstrated that existing online resources were generally of poor quality and lacked important content. With this knowledge, we created a LARS educational booklet and developed an online app containing LARS educational material and an interactive forum for online peer support. We are now in an optimal position to rigorously test the potential effects of this initiative on patient-centered outcomes.

This study is a multicenter, randomized, assessor-blind, parallel-groups, pragmatic trial involving patients from 5 large colorectal surgery practices (Jewish General Hospital, McGill University Health Centre-Montreal, QC; Toronto Western Hospital, Mount Sinai Hospital- Toronto, ON; Saint Paul's Hospital-Vancouver, BC). Participants will be randomized into the intervention group, who will have access to the online peer support app, and the control group who will only receive a LARS patient educational booklet. Trained peer support mentors will moderate discussion in the peer support forum, which will also be monitored daily by expert health care professionals. Data regarding patient demographics, disease and treatment characteristics will be obtained via hospital chart review. The primary outcome will be health- related quality of life at 6 months. Secondary outcomes will be patient activation and bowel function. We hypothesize that availability of this app (consisting of LARS information, a closed forum for discussion among peers and trained peer support mentors) improves health-related quality of life when compared to the comparison group.

Given the significant numbers of patients who suffer from LARS symptoms following restorative proctectomy and the potential chronic nature of their symptoms, this RCT has the potential to contribute important knowledge to support patient-centered care of rectal cancer survivors. The technology addressed in this study (a mobile app for information and online peer support) is readily accessible and can be relatively easily implemented across large range of geographic jurisdictions and surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* underwent restorative protectomy for Neo-plastic disease of the rectum
* completed all treatment within the last 3 years
* patients with minor or major LARS as defined with the LARS score.

Exclusion Criteria:

* Active chemotherapy or radiotherapy
* Major colonic resection in addition to protectomy
* Cannot be contacted by telephone
* Unable to read and comprehend English/French
* Does not have the appropriate interface to access the app
* Unable to give clear and informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire - C30 questionnaire | 1 week before the launch of the app
  Questionnaire measures baseline quality of life before app use. Maximum score 100 (better function, quality of life). Minimum score 0 (worse function, quality of life).
Assessing 'Change' via European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire - C30 questionnaire after 6 months | 6 months after using the app.
  Questionnaire measures change in quality of life after app use. Maximum score 100 (better function, quality of life). Minimum score 0 (worse function, quality of life).

SECONDARY OUTCOMES:
Patient activation measures | 1 week before the launch of the app
  Questionnaire measures patient activation before app use. Maximum score 52 (higher patient activation), Minimum score 13 (lower patient activation).
Change in Patient activation measures | 6 months after using the app.
  Questionnaire measures patient activation after app use. Maximum score 52 (higher patient activation), Minimum score 13 (lower patient activation).
Bowel function Low Anterior Resection Syndrome score | 1 week before the launch of the app
  Questionnaire measures bowel function before app use. Maximum score 42 (worse bowel function). Minimum score 0 (better bowel function)
Bowel function Low Anterior Resection Syndrome score | 6 months after using the app.
  Questionnaire measures bowel function after app use. Maximum score 42 (worse bowel function). Minimum score 0 (better bowel function)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - St Paul's Hospital, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No